CLINICAL TRIAL: NCT01968460
Title: A Phase 2B, Twelve-week Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study, To Determine the Safety, Tolerability and Efficacy of Two Doses of Once Daily P2B001 in Subjects With Early Parkinson's Disease
Brief Title: Safety, Tolerability and Efficacy of Two Doses of Once Daily P2B001 in Subjects With Early Parkinson's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pharma Two B Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P2B001/001
Record Dates: First submitted 2013-10-15; First posted 2013-10-24 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2015-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease, Rasagiline, Pramipexole
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole; rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- P2B001 once daily (pramipexole 0.6 mg / rasagiline 0.75 mg), (Experimental): Fixed Dose Combination of pramipexole 0.6 mg and rasagiline 0.75 mg once daily.
  Interventions: Drug: P2B001 once daily (pramipexole 0.6 mg / rasagiline 0.75 mg),
- P2B001 once daily (pramipexole 0.3 mg / rasagiline 0.75 mg), (Experimental): Fixed Dose Combination of pramipexole 0.3 mg and rasagiline 0.75 mg once daily
  Interventions: Drug: P2B001 once daily (pramipexole 0.3 mg / rasagiline 0.75 mg),
- Placebo (Placebo Comparator): Placebo once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P2B001 once daily (pramipexole 0.6 mg / rasagiline 0.75 mg), — Fixed Dose Combination of pramipexole 0.6 mg and rasagiline 0.75 mg once daily
  Arms: P2B001 once daily (pramipexole 0.6 mg / rasagiline 0.75 mg),
Drug: Placebo — placebo
  Arms: Placebo
Drug: P2B001 once daily (pramipexole 0.3 mg / rasagiline 0.75 mg), — Fixed Dose Combination of pramipexole 0.3 mg and rasagiline 0.75 mg once daily
  Arms: P2B001 once daily (pramipexole 0.3 mg / rasagiline 0.75 mg),

SUMMARY:
This study will evaluate an oral fixed-dose, once daily product that combines pramipexole and rasagiline for the treatment of early Parkinson's disease.

Animal studies support the therapeutic advantage of combining low doses of rasagiline and pramipexole and suggest further improvement when both are administered in a sustained fashion. Both rasagiline and pramipexole are well known marketed drugs for Parkinson's disease with a good safety profile. combining the drugs in low doses and controlled release may provide better symptom management than the existing drugs alone or together.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female ≥35 years of age to ≤75 years of age at the time of enrollment.
* Subject has idiopathic Parkinson's disease consistent with the UK Brain Bank Criteria; must have bradykinesia with sequence effect and rest tremor or prominent motor asymmetry.
* Subject with disease duration no longer than 3 years and 0 months.
* Subject has a Hoehn & Yahr (H&Y) stage score of < 3.
* Subject has a MMSE score ≥ 26

Exclusion Criteria:

* Subject has an atypical parkinsonian syndrome or secondary parkinsonism (e.g., due to drugs, metabolic neurogenetic disorders, encephalitis, cerebrovascular disease or degenerative disease).
* Subject has a history of psychosis or hallucinations within the previous 12 months.
* Subject who is taking anticholinergic drugs.
* Subject has previous exposure to levodopa or a dopamine agonist for longer than 4 weeks; if previous exposure was less than 4 weeks then it must not be within 2 months prior to the baseline visit.
* Subject has previous exposure to a MAO-B inhibitor for longer than 4 weeks; if previous exposure was less than 4 weeks then it must not be within 3 months prior to the baseline visit.
* Subject who is taking MAO inhibitors, potent CYP1A2 inhibitors, e,g, Ciprofloxacin, Dextromethorphan or antitussive agent, analgesic agents such as tramadol, meperidine, methadone and propoxyphene, strong 3A4 inducers, e.g., St. John's Wort or cyclobenzaprine (tricyclic muscle relaxant), dopamine antagonists, such as the neuroleptics (phenothiazines, butyrophenones, thioxanthenes) or metoclopramide. Probenecid, cimetidine, ranitidine, diltiazem, verapamil and quinidine.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: pninit litman, Ph.D, Study Director — Pharma Two B Ltd.
Locations (29):
- United States (24):
  - P2B001 Site Birmingham, Birmingham, Alabama
  - P2B001 Site Los Angeles, Los Angeles, California
  - P2B001 Site Aurora, Aurora, Colorado
  - P2B001 Manchester, Manchester, Connecticut
  - P2B001 Site New Haven, New Haven, Connecticut
  - P2B001 Site Boca Raton, Boca Raton, Florida
  - P2B001 Site Port Charlotte, Port Charlotte, Florida
  - P2B001 Site Tampa, Tampa, Florida
  - P2B001 Site Augusta, Augusta, Georgia
  - P2B001 site Chicago, Chicago, Illinois
  - P2B001 Site Kansas City, Kansas City, Kansas
  - P2B001 Site Boston, Boston, Massachusetts
  - P2B001 Site west Bloomfield, West Bloomfield, Michigan
  - P2B001 Site Golden Valley, Golden Valley, Minnesota
  - P2B001 Site Camden, Camden, New Jersey
  - P2B001 Site New Brunswick, New Brunswick, New Jersey
  - P2B001 site Commack, Commack, New York
  - P2B001 Site New York, New York, New York
  - P2B001 Site Durham, Durham, North Carolina
  - P2B001 Site Cincinnati, Cincinnati, Ohio
  - P2B001 Site Toledo, Toledo, Ohio
  - P2B001 Site Tulsa, Tulsa, Oklahoma
  - P2B001 Site Houston, Houston, Texas
  - P2B001 Site Roanoke, Roanoke, Virginia
- Israel (5):
  - P2B001 Site Rambam Israel, Haifa
  - P2B001 Site Belinson, Pethch Tikva
  - P2B001 Site Sheba Medical Center, Ramat Gan
  - P2B001 Site Asaf Harofe, Rishon LeZiyyon
  - P2B001 Site Sourasky Medical Center, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- P2B001 Treatment A: Fixed Dose Combination of pramipexole 0.6 mg and rasagiline 0.75 mg once daily.
  P2B001 once daily (pramipexole 0.6 mg / rasagiline 0.75 mg), : Fixed Dose Combination of pramipexole 0.6 mg and rasagiline 0.75 mg once daily
- P2B001 Treatment B: Fixed Dose Combination of pramipexole 0.3 mg and rasagiline 0.75 mg once daily
  P2B001 once daily (pramipexole 0.3 mg / rasagiline 0.75 mg), : Fixed Dose Combination of pramipexole 0.3 mg and rasagiline 0.75 mg once daily
Period: Overall Study
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo
Started | 49 | 50 | 50
Completed | 43 | 45 | 48
Not Completed | 6 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo | Total
Number analyzed (Participants) | 49 | 50 | 50 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 18 | 66
  >=65 years | 24 | 27 | 32 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 63 (8) | 64 (7) | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 19 | 49
  Male | 35 | 34 | 31 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 1 | 8
  White | 46 | 43 | 47 | 136
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 42 | 126
  Israel | 7 | 8 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Total UPDRS I, II, III Scores
Description: Change from baseline to final visit (week 12) in total UPDRS score (defined as sum of parts I, II and III, scores (0-176). UPDRS- Unified Parkinson's Disease Rating Scale, minimum value is 0 points and maximum value is 176.
  High score mean worse outcome.
Time Frame: Week 12
Population: ITT analyis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo
Number analyzed (Participants) | 49 | 50 | 50
units on a scale | -5.97 (0.94) | -5.15 (0.9) | -1.31 (0.88)
Statistical Analysis 1: Comparison: P2B001 Treatment A vs Placebo; Test type: Superiority; p = 0.0004, MMRM — The overall significance level for this study will be 5% using two-tailed tests utilizing the hierarchical gate keeping approach to control the overall Type-I error rate in the strong sense; Mean Difference (Net) = -4.67, 95% CI 2-sided [-7.20 to -2.13], Standard Error of Mean 1.28
Statistical Analysis 2: Comparison: P2B001 Treatment B vs Placebo; Test type: Superiority; p = 0.0027, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.84, 95% CI 2-sided [-6.32 to -1.36], Standard Error of Mean 1.25

2. Secondary Outcome: UPDRS ADL (Part II)
Description: Change from baseline in individual UPDRS ADL (part II). Activity of daily Life UPDRS part II minimum is 0 point and max is 52 point (worse outcome)
Time Frame: Week 12
Population: ITT analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo
Number analyzed (Participants) | 49 | 50 | 50
units on a scale | -1.49 (0.37) | -1.06 (0.36) | 0.36 (0.39)
Statistical Analysis 1: Comparison: P2B001 Treatment A vs Placebo; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.85, 95% CI 2-sided [-2.86 to -0.84], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: P2B001 Treatment B vs Placebo; Test type: Superiority; p = 0.005, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.42, 95% CI 2-sided [-2.41 to 0.44], Standard Error of Mean 0.01

3. Secondary Outcome: CGI-S
Description: Change from baseline in individual Clinical Global Impression - Severity. Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness (Parkinson's Disease) at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis as one of the following:. 1 is normal and 7 is the most extremely ill patients. A subject defined as a treatment responder when the improvement from baseline to the Week12 / Last Observed Value (LOV) was of at least 1 point or more.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo
Number analyzed (Participants) | 49 | 50 | 50
Participants | 13 | 9 | 3
Statistical Analysis 1: Comparison: P2B001 Treatment A vs Placebo; A subject will be defined as a treatment responder in case that the improvement from baseline to the Week12 / Last Observed Value (LOV) in the CGI-S will be of 1 point or more. Baseline adjusted logistic regression (SAS® LOGISTIC procedure) stratified by GeoSite using the STRATA sub-command with the following effects: treatment group and baseline CGI-S measurement was used to test the between the active groups and placebo contrasts; Test type: Superiority; p = 0.0165, Regression, Logistic — The overall significance level for this study was 5% using two-tailed tests; Odds Ratio (OR) = 8.10, 95% CI 2-sided [1.47 to 44.77]
Statistical Analysis 2: Comparison: P2B001 Treatment B vs Placebo; Test type: Superiority; p = 0.111, Regression, Logistic — The overall significance level for this study will be 5% using two-tailed tests; Odds Ratio (OR) = 4.23, 95% CI 2-sided [0.72 to 24.90], Standard Error of Mean 0.90

4. Secondary Outcome: UPDRS Motor (Part III)
Description: Change from baseline in individual UPDRS motor (part III). UPDRS- Unified Parkinson's Disease Rating Scale, part III motor . min is 0 and Max is 108 (Worse outcome)
Time Frame: 12 weeks
Population: ITT anlysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo
Number analyzed (Participants) | 49 | 50 | 50
units on a scale | -4.43 (0.74) | -3.95 (0.7) | -1.62 (0.69)
Statistical Analysis 1: Comparison: P2B001 Treatment A vs Placebo; Test type: Superiority; p = 0.0058, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.81, 95% CI 2-sided [-4.80 to -0.83], Standard Error of Mean 1.00
Statistical Analysis 2: Comparison: P2B001 Treatment B vs Placebo; Test type: Superiority; p = 0.0191, MMRM — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.32, 95% CI 2-sided [-4.26 to -0.39], Standard Error of Mean 0.98

5. Secondary Outcome: PDQ39
Description: Change from baseline in individual Parkinson's Disease Questionnaire - 39. Score 0-100 where 0 is indicative of no problem at all and 100 is the maximum level of problem.
Time Frame: 12 weeks
Population: ITT Analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo
Number analyzed (Participants) | 49 | 50 | 50
units on a scale | -3.01 (0.89) | -2.19 (0.88) | 0.26 (0.88)
Statistical Analysis 1: Comparison: P2B001 Treatment A vs Placebo; Test type: Superiority; p = 0.0097, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.27, 95% CI 2-sided [-5.72 to -0.80], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: P2B001 Treatment B vs Placebo; Test type: Superiority; p = 0.0509, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.45, 95% CI 2-sided [-4.91 to -0.012], Standard Error of Mean 1.24

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | P2B001 Treatment A | P2B001 Treatment B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 37/49 | 20/50 | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P2B001 Treatment A (N=49) | P2B001 Treatment B (N=50) | Placebo (N=50)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — NON-ST ELEVATION MYOCARDIAL INFARCTION
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P2B001 Treatment A (N=49) | P2B001 Treatment B (N=50) | Placebo (N=50)
NAUSEA (Gastrointestinal disorders) | 10 (12) | 6 (6) | 1 (1) — NAUSEA
SOMNOLENCE (Nervous system disorders) | 8 (9) | 4 (5) | 0 (0) — SOMNOLENCE
DIZZINESS (Nervous system disorders) | 5 (6) | 2 (2) | 4 (4) — DIZZINESS
fatigue (General disorders) | 4 (4) | 1 (1) | 1 (1)
nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 5 (6)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
tremor (Nervous system disorders) | 4 (5) | 3 (3) | 3 (3)
insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2)
orthostatic hypotension (Vascular disorders) | 2 (3) | 1 (1) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No